CLINICAL TRIAL: NCT06872671
Title: The Effect of Breathing Exercises and the Valsalva Maneuver on Pain Reduction During Peripheral Intravenous Catheterization: A Randomized Controlled Trial
Brief Title: The Effect of Breathing Exercises and the Valsalva Maneuver on Pain Reduction During Peripheral Intravenous Catheterization
Acronym: Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Sumeyye Akcoban, Principal Investigator, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMKU-KMY-SA-03
Record Dates: First submitted 2025-02-28; First posted 2025-03-12 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Pain
Keywords: pain; nursing; breathing exercises; valsalva maneuver
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Parallel 3 group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breathing Exercise Group (Experimental): After patients receive training on the breathing exercise, nurses responsible for performing the PIVC procedure will be provided with the necessary information regarding the intervention. It will be emphasized that patients should begin the breathing exercise before the PIVC procedure. Additionally, nurses will be instructed to perform the catheterization during the fifth step of the breathing exercise.
  Before the PIVC procedure in the breathing exercise group, the researcher will be present alongside the nurse performing the intervention. Nurses will be informed that they should initiate the PIVC procedure three seconds after the patient reaches the fourth step, which involves breath-holding. Furthermore, efforts will be made to ensure that the same nurse performs the PIVC procedure for each patient in the breathing exercise group.
  Hemodynamic variables, including blood pressure, pulse rate, and oxygen saturation, will be recorded before and after the breathing exercise.
  Interventions: Other: Experimental: Breathing Exercise Group
- Valsalva Manoeuvre Group (Experimental): Care will be taken to ensure that the PIC procedure is performed by the same nurse for the patients in the Valsalva manoeuvre group. The nurses performing the PIC procedure will be informed about the subject of the research and will be told that the patients will start the valsalva manoeuvre before the PIC procedure. Patients who can perform the valsalva manoeuvre by the researcher will be included in the study. Haemodynamic variables (blood pressure, pulse, saturation) of the patients will be recorded before the application of the Valsalva manoeuvre. Afterwards, the researcher will instruct the patients to blow into the plastic tube for 20 seconds after a deep breath to create 30 mmHg pressure. After the application of the Valsalva manoeuvre, haemodynamic variables (blood pressure, pulse, saturation) of the patients will be recorded.
  Interventions: Other: Valsalva Manoeuvre Group
- Control Group (No Intervention): In the control group, the routine PIVC procedure will be performed by the same nurse for all patients. No additional interventions will be applied. Each patient's pain will be assessed and recorded before, during, and after the PIVC procedure by an independent nurse who is not involved in the study.

INTERVENTIONS:
Other: Experimental: Breathing Exercise Group — Eyes will be closed first. Head and neck will be relaxed. Breathing will be taken through the nose for three seconds. Then the breath will be held for three seconds. In the last step, breath will be exhaled through the mouth for three seconds. The patient will be instructed to take five normal breaths between each breathing exercise. The patient will be asked to count to three and will be told that he/she can count by using his/her fingers. The exercise will be started two minutes before the catheterisation procedure and the patient will be instructed to perform the breathing exercise twice. The patient will be asked to continue doing the breathing exercise until the PIC application process is completed.
  Arms: Breathing Exercise Group
Other: Valsalva Manoeuvre Group — The valsalva manoeuvre will be performed by blowing into a plastic tube connected through a sphygmomanometer. Patients will be allowed to raise the manometer by 30 mmHg for at least 20 seconds. Care will be taken to ensure that the PIC procedure is performed by the same nurse for the patients in the Valsalva manoeuvre group. The nurses performing the PIC procedure will be informed about the research subject and will be told that the patients will start the valsalva manoeuvre before the PIC procedure. Patients who can perform the valsalva manoeuvre by the researcher will be included in the study. Haemodynamic variables (blood pressure, pulse, saturation) of the patients will be recorded before the valsalva manoeuvre. Afterwards, the researcher will instruct the patients to blow into the plastic tube for 20 seconds after a deep breath to create 30 mmHg pressure.
  Arms: Valsalva Manoeuvre Group

SUMMARY:
Peripheral intravenous catheter (PIVC) insertion is a painful procedure due to its invasive nature. During the procedure, damage to the endothelial layer and improper interventions can further increase pain levels. Additionally, pain can cause vasoconstriction, negatively affecting venous filling and reducing the success rate of IV catheter insertion. Both pharmacological and non-pharmacological methods are used to alleviate invasive pain associated with PIVC. However, pharmacological methods are often considered disadvantageous due to their high cost, potential adverse effects, and increased medication use. In contrast, non-pharmacological approaches are preferred as they are cost-effective, have fewer side effects, and pose a lower risk of complications.

DETAILED DESCRIPTION:
One of the non-pharmacological methods used for pain reduction is breathing exercises. As a distraction technique, breathing exercises have been increasingly utilized to alleviate invasive pain experienced during blood collection and cannulation procedures. By enhancing lung ventilation, deep breathing maximizes oxygen intake, leading to relaxation in the patient. This state of relaxation contributes to a sense of comfort and reduces the perception of pain.

A review of the literature revealed only one study specifically evaluating the effectiveness of breathing exercises in reducing pain during PIVC insertion. Existing research has reported that breathing exercises have a positive impact on pain experienced during PIVC placement. In these studies, individuals were first positioned comfortably. They were then instructed to take a slow, deep breath through the nose, hold it briefly, and exhale slowly through the mouth. During inhalation, participants were guided to expand their abdomen and push the diaphragm downward, while during exhalation, they were asked to contract the abdominal muscles, draw the abdomen inward, and push the diaphragm upward. Additionally, individuals were instructed to silently count to four while inhaling, holding their breath, and exhaling. The breathing exercise began one minute before the procedure and continued throughout its duration.

Another non-pharmacological method used for pain reduction is the Valsalva maneuver, a well-known breathing technique. The Valsalva maneuver involves a forceful exhalation against a closed airway, stimulating the vagus nerve and causing physiological changes, particularly in heart rate and blood pressure. These physiological effects make the Valsalva maneuver a valuable diagnostic and therapeutic tool for terminating supraventricular tachycardia, assessing cardiac murmurs and left ventricular function, managing neuropathy, and controlling pain.

A review of the literature identified a few studies evaluating the effects of the Valsalva maneuver on pain, anxiety, and vital signs during PIVC insertion. The findings of these studies indicate that the Valsalva maneuver has a positive effect in reducing pain experienced during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years of age or older,

  * Hospitalised in the general surgery ward with PIC indication,
  * Non-users of central nervous system drugs,
  * No heart and lung disease,
  * Absence of phlebitis, scar tissue, dermatitis, incision and infection in the area to be accessed,
  * No analgesic or anaesthetic agent has been administered 24 hours prior to PIC administration,
  * No pain in any part of the body that may affect the results of the study,
  * No PIK experience in the last month, The one with the -20-G catheter,
  * Pressure pain threshold averages 8-16 pounds (Lb),
  * No communication problems,
  * Capable of breathing exercise practice,
  * No mental problems,
  * Patients who agree to participate in the study will be included.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Patient Identification Information Form | up to 12 weeks
  A descriptive information form was created by examining the studies with patients who underwent peripheral intravenous catheterisation. In the descriptive information form; 6 questions including the patient's age, height, weight, pressure pain threshold value and haemodynamic indicators (blood pressure, pulse, saturation) were asked.
Baseline Algometer (66 Lb/30 Kg) | up to 12 weeks
  Algometer is a widely used device for determining pressure pain threshold measurements. Pressure pain threshold can be defined as the minimum force applied to elicit pain. The measurement assessed with a pressure algometer is a manual procedure that requires a perceptual response from the individual. In order to introduce the Baseline Algometer (66 Lb/30 Kg) tool to the patients who are considered to be included in the study, pressure will be applied to a different area (above the wrist) outside the area to be measured. Patients will be asked to give the "stop" command at the first sensation of pain and the application will be repeated 3 times in all patients to ensure that the patients adapt to the real application. Then, the mean pressure pain threshold will be determined after three measurements made at 5-second intervals from the right antecubital region of the patients. Patients with an average pressure pain threshold of 8-16 pounds
Visual Comparison Scale | up to 12 weeks
  The Turkish validity and reliability of this scale developed by Price et al. (1994) to evaluate the severity of pain was performed by Eti Aslan (2004) by evaluating the presence of pain in patients in the postoperative period. The scale is graded from 0 to 10, where 0 = no pain and 10 = unbearable pain. The severity of pain before, during (during peripheral intravenous catheterisation) and after PIC application will be recorded by a nurse independent of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yilmaz D, Gunes UY. The effect on pain of three different nonpharmacological methods in peripheral intravenous catheterisation in adults. J Clin Nurs. 2018 Mar;27(5-6):1073-1080. doi: 10.1111/jocn.14133. Epub 2018 Jan 8. PMID 29076581
- [Result] Ozkan O, Korkut S. Effect of Breathing Exercise During Peripheral Venous Catheterization on Pain, Anxiety, and Patient Satisfaction: A Randomized Controlled Trial. J Perianesth Nurs. 2024 Aug;39(4):630-637. doi: 10.1016/j.jopan.2023.11.006. Epub 2024 Feb 29. PMID 38430076
- [Derived] Akcoban S, Tosun B. Breathing Exercises, Valsalva Maneuver Reduce Pain in Peripheral Intravenous Catheterization: Randomized Trial. Pain Manag Nurs. 2025 Nov 21:S1524-9042(25)00301-7. doi: 10.1016/j.pmn.2025.10.010. Online ahead of print. PMID 41274790